CLINICAL TRIAL: NCT06901856
Title: Modified Cap-assisted Endoscopic Mucosal Resection and Modified Endoscopic Mucosal Resection with a Ligation Device for Small Rectal Neuroendocrine Tumors Less Than 1 Cm: a Muticenter Randomized Noninferiority Trial
Brief Title: Endoscopic Resection for Small Rectal Neuroendocrine Tumors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025-063-02
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Rectal Neuroendocrine Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mEMR-C group (Experimental): In mEMR-C group, enrolled patients will receive modified EMR-C without submucosal injection.
  Interventions: Procedure: mEMR-C procedure
- mEMR-L group (Active Comparator): In mEMR-L group, enrolled patients will receive modified ESMR-L without submucosal injection.
  Interventions: Procedure: mEMR-L procedure

INTERVENTIONS:
Procedure: mEMR-C procedure — A transparent cap with an inner groove (MH-593; Olympus, Tokyo, Japan) was attached to the forward-viewing colonoscope. After the endoscope was inserted into the rectum, a crescent-shaped electrosurgical snare was passed through the sheath and looped along the inner groove of the cap. Submucosal injections were not required in this method. The tumor was suctioned into the cap and grasped by tightening the snare. After confirming the appropriate snare placement, both the tumor and overlying mucosa were resected using electric cautery (Endocut Q, effect 2, VIO 200D; ERBE, Tübingen, Germany), and the resected tumor was sent for pathological examination. Endoscopic examination was repeated without a transparent cap to evaluate the wound carefully in cases of perforation or bleeding and to ensure the absence of residual tumor tissues. If there was spurting or active bleeding, hot forceps were used to stop the bleeding.
  Arms: mEMR-C group
Procedure: mEMR-L procedure — First, install the ligation device (provided by Jiangsu Gerrit) at the front end of the endoscope. After inserting the endoscope into the rectum, suck the lesion into the ligation device, release the ligator to ligate the lesion. Then, use a snare to resect the lesion below the ligator. Finally, uniformly suture the wound surface with metal clips.
  Arms: mEMR-L group

SUMMARY:
According to clinical practice and relevant retrospective research data, both modified cap-assisted endoscopic mucosal resection (mEMR-C) and endoscopic mucosal resection with a ligation device(ESMR-L) were reported to be effective for the treatment of small rectal neuroendocrine tumors (NETs) . However, there is a lack of multicenter prospective studies to evaluate the advantages and disadvantages of mEMR-C and mEMR-L. mEMR-C is the modified ESMR-L without submucosal injection.

DETAILED DESCRIPTION:
We aimed to conduct a muticenter randomized controlled trial to compare mEMR-C with mEMR-L for the treatment of small rectal neuroendocrine tumors (NETs) in ten tertiary hospitals in China.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 80 years;
2. With a high suspicion or evidence of rectal NET assessed using EUS or colonoscopy;
3. With tumor size ≤10 mm assessed by colonoscopy;
4. Plan to receive mEMR-C or mEMR-L treatment and provide written informed consent;

Exclusion Criteria:

1. Unable to tolerate mEMR-L or mEMR-C as assessed by the research team of each center;
2. Complicated with serious diseases such as malignant tumor, which may lead to shorter life expectancy, the research team considers that it is not suitable for inclusion in the study after comprehensive evaluation;
3. Rectal NET with lymph node metastasis or distant metastasis;
4. Received resection of rectal neuroendocrine tumor by other surgical procedures;
5. Multiple rectal neuroendocrine tumors;
6. Vulnerable groups such as pregnant women or patients with mental disorders;
7. Poor compliance, unable to cooperate with treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
histological complete resection | within 14 days after procedure
  complete single-piece (en bloc) resection of the targeted lesion with horizontal and vertical free margins.

SECONDARY OUTCOMES:
success rate of operation | intraoperative
  the proportion of patients whose tumors were successfully resected in each group
en bloc resection | intraoperative
  complete single resection of the targeted lesion, irrespective of whether the basal and lateral tumor margins were infiltrated or undetermined
operation time | intraoperative
  the time required to complete the procedure, was taken from the installation of the snare in the mEMR-C or the first submucosal injection in ESD to the end of complete resection of the targeted area or a failure or complication of the procedure which required discontinuation
complications | within 14 days after procedure
  perforation or hemorrhage during or after operation
length of stay | within 14 days after procedure
  calculated from the day of admission to day of discharge
hospitalization cost | within 14 days after procedure
  represent the hospital's costs of being hospitalized
operation cost | within 14 days after procedure
  the cost of mEMR-C or mEMR-L procedures, except the cost of other endoscopic procedures
histopathologic grade | within 14 days after procedure
  NET grade 1, NET grade 2, NET grade 3, and NEC